CLINICAL TRIAL: NCT04622137
Title: An Alternative Conservative Treatment Method For Midshaft Clavicular Fractures: Kinesiotaping Therapy
Brief Title: Kinesiotaping Therapy for Clavicular Fractures FRACTURES:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist,Chief assistant, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kinesiotaping Therapy
Record Dates: First submitted 2020-10-15; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Clavicle Fracture
Keywords: kinesiotherapy; arm sling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm sling only group (group S) (No Intervention): Participants used only arm sling for clavicula fracture
- Arm sling with kinesiotaping therapy group (group K). (Active Comparator): Participants used arm sling and the investigators applied kinesiotheraphy for clavicula fracture
  Interventions: Procedure: Kinesiotaping therapy

INTERVENTIONS:
Procedure: Kinesiotaping therapy — The investigators used kinesiotaping strips in formations such as the Y, I, X, fan, web, and donut formations ove fractured clavicula.
  Arms: Arm sling with kinesiotaping therapy group (group K).

SUMMARY:
This is a multicenter prospective randomized controlled study. Forty patients in whom conservative treatment for clavicle midshaft fractures was indicated between January 2018 and July 2019 were included.

The investigators aimed to evaluate the effectiveness of the kinesiotaping technique for the conservative treatment of clavicle midshaft fractures. The investigators hypothesized that kinesiotaping reduces the disadvantages of conservative treatment, such as early-phase pain, high nonunion rates, and a prolonged time to return to work, and yields better clinical and functional outcomes by providing good mechanical support and neutralizing the deforming muscle forces around the fractured clavicle.

DETAILED DESCRIPTION:
The investigators divided into 2 groups and followed one group of patients with clavicle fractures only with shoulder sling, while the other group were followed with kinesiotherapy treatment and shoulder arm sling. They investigated the effect of kinesiotherapy treatment on early pain and returning time to work.

ELIGIBILITY:
Inclusion Criteria:

Participants with midclavicle fracture within 24 hours

Exclusion Criteria:

Participants with open fractures,

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the two groups in terms of early return to work | 6. months
  The investigators aim is to examine the effect of kinesiotaping treatment on clavicle fracture union.

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Qin M, Zhao S, Guo W, Tang L, Li H, Wang X, Zhu Z, Sun T. Open reduction and plate fixation compared with non-surgical treatment for displaced midshaft clavicle fracture: A meta-analysis of randomized clinical trials. Medicine (Baltimore). 2019 May;98(20):e15638. doi: 10.1097/MD.0000000000015638. PMID 31096481
- [Background] Sang QH, Gou ZG, Zheng HY, Yuan JT, Zhao JW, He HY, Liu C, Liu Z. The Treatment of Mid-shaft Clavicle Fractures. Chin Med J (Engl). 2015 Nov 5;128(21):2946-51. doi: 10.4103/0366-6999.168068. PMID 26521795
- [Background] Craig EV. Fractures of the Clavicle. In: Rockwood CA, Green DP, Bucholz RW, Heckman JD, Editors. Rockwood and Green's Fractures in Adults. Philadelphia, PA: Lippincott- Raven; 1996. p. 1109-1161.
- [Background] Tamaoki MJS, Matsunaga FT, Costa ARFD, Netto NA, Matsumoto MH, Belloti JC. Treatment of Displaced Midshaft Clavicle Fractures: Figure-of-Eight Harness Versus Anterior Plate Osteosynthesis: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Jul 19;99(14):1159-1165. doi: 10.2106/JBJS.16.01184. PMID 28719554
- [Background] Jones GL, Bishop JY, Lewis B, Pedroza AD; MOON Shoulder Group. Intraobserver and interobserver agreement in the classification and treatment of midshaft clavicle fractures. Am J Sports Med. 2014 May;42(5):1176-81. doi: 10.1177/0363546514523926. Epub 2014 Feb 26. PMID 24573571
- [Background] Wiesel B, Nagda S, Mehta S, Churchill R. Management of Midshaft Clavicle Fractures in Adults. J Am Acad Orthop Surg. 2018 Nov 15;26(22):e468-e476. doi: 10.5435/JAAOS-D-17-00442. PMID 30180095
- [Background] Ersen A, Atalar AC, Birisik F, Saglam Y, Demirhan M. Comparison of simple arm sling and figure of eight clavicular bandage for midshaft clavicular fractures: a randomised controlled study. Bone Joint J. 2015 Nov;97-B(11):1562-5. doi: 10.1302/0301-620X.97B11.35588. PMID 26530661
- [Background] Hill JM, McGuire MH, Crosby LA. Closed treatment of displaced middle-third fractures of the clavicle gives poor results. J Bone Joint Surg Br. 1997 Jul;79(4):537-9. doi: 10.1302/0301-620x.79b4.7529. PMID 9250733
- [Background] Kaplan S, Alpayci M, Karaman E, Cetin O, Ozkan Y, Ilter S, Sah V, Sahin HG. Short-Term Effects of Kinesio Taping in Women with Pregnancy-Related Low Back Pain: A Randomized Controlled Clinical Trial. Med Sci Monit. 2016 Apr 18;22:1297-301. doi: 10.12659/msm.898353. PMID 27088271
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Akca AH, Sasmaz MI, Kaplan S. Kinesiotaping for isolated rib fractures in emergency department. Am J Emerg Med. 2020 Mar;38(3):638-640. doi: 10.1016/j.ajem.2019.11.049. Epub 2019 Dec 20. PMID 31937442
- [Background] Alexander CM, Stynes S, Thomas A, Lewis J, Harrison PJ. Does tape facilitate or inhibit the lower fibres of trapezius? Man Ther. 2003 Feb;8(1):37-41. doi: 10.1054/math.2002.0485. PMID 12586560
- [Background] Schemitsch LA, Schemitsch EH, Veillette C, Zdero R, McKee MD. Function plateaus by one year in patients with surgically treated displaced midshaft clavicle fractures. Clin Orthop Relat Res. 2011 Dec;469(12):3351-5. doi: 10.1007/s11999-011-1915-x. PMID 21590485
- [Background] Stanley D, Trowbridge EA, Norris SH. The mechanism of clavicular fracture. A clinical and biomechanical analysis. J Bone Joint Surg Br. 1988 May;70(3):461-4. doi: 10.1302/0301-620X.70B3.3372571.
- [Background] Naveen BM, Joshi GR, Harikrishnan B. Management of mid-shaft clavicular fractures: comparison between non-operative treatment and plate fixation in 60 patients. Strategies Trauma Limb Reconstr. 2017 Apr;12(1):11-18. doi: 10.1007/s11751-016-0272-4. Epub 2017 Jan 4. PMID 28054249
- [Background] Caglar A, Pekyavas NO, Tigli AA, Aytar A, Baltaci G. Are the Kinesio Tape colors effective for patient perception? A randomized single blind trial. J Exerc Ther Rehabil 2016;3:96-101.
- [Background] Woltz S, Krijnen P, Schipper IB. Plate Fixation Versus Nonoperative Treatment for Displaced Midshaft Clavicular Fractures: A Meta-Analysis of Randomized Controlled Trials. J Bone Joint Surg Am. 2017 Jun 21;99(12):1051-1057. doi: 10.2106/JBJS.16.01068. PMID 28632595
- [Background] Burnham JM, Kim DC, Kamineni S. Midshaft Clavicle Fractures: A Critical Review. Orthopedics. 2016 Sep 1;39(5):e814-21. doi: 10.3928/01477447-20160517-06. Epub 2016 May 25. PMID 27220117
- [Background] Postacchini F, Gumina S, De Santis P, Albo F. Epidemiology of clavicle fractures. J Shoulder Elbow Surg. 2002 Sep-Oct;11(5):452-6. doi: 10.1067/mse.2002.126613. PMID 12378163
- [Background] Thormodsgard TM, Stone K, Ciraulo DL, Camuso MR, Desjardins S. An assessment of patient satisfaction with nonoperative management of clavicular fractures using the disabilities of the arm, shoulder and hand outcome measure. J Trauma. 2011 Nov;71(5):1126-9. doi: 10.1097/TA.0b013e3182396541. PMID 22071918
- [Background] Kase K, Wallis J, Kase T. Clinical Therapeutic Applications of the Kinesio Taping® Method. Dallas, TX: Kinesio Taping Association; 2003.
- [Background] Waldmann S, Benninger E, Meier C. Nonoperative Treatment of Midshaft Clavicle Fractures in Adults. Open Orthop J. 2018 Jan 17;12:1-6. doi: 10.2174/1874325001812010001. eCollection 2018. PMID 29430265
- [Background] Figueiredo GS, Tamaoki MJ, Dragone B, Utino AY, Netto NA, Matsumoto MH, Matsunaga FT. Correlation of the degree of clavicle shortening after non-surgical treatment of midshaft fractures with upper limb function. BMC Musculoskelet Disord. 2015 Jun 17;16:151. doi: 10.1186/s12891-015-0585-3. PMID 26080806